CLINICAL TRIAL: NCT01399177
Title: Influence of Changes in Food Group Variety on Food Cravings, Energy Intake, and Weight Loss After Bariatric Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Other Study IDs: 3177
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to find out if there is any change in diet on food cravings and weight loss in the 12 months following bariatric surgery.

DETAILED DESCRIPTION:
Research suggests that satiation processes in obese patients may be impaired, possibly resulting in excessive energy intake and poorer weight loss outcomes. One factor that may contribute to disruption of satiation processes and related overconsumption is dietary variety. Additionally, food cravings for restricted foods are believed to contribute to poor compliance to diets, and in controlled feeding studies, food cravings are the most frequently provided reason for poor dietary adherence. Interestingly, several investigations have found that cravings decrease when individuals follow a very-low-calorie or monotonous diet (9-11). Thus, reductions in the variety of the diet may also reduce food cravings, and assist in dietary adherence. It is also possible that the type of surgical procedure performed may influence changes in dietary variety, and consequently food cravings. To date, few studies have analyzed bariatric surgery patients' selection of foods within specific food groups and no study has examined the variety of foods consumed within food groups. Changes in food group variety which facilitate improvements in regulation of energy intake and body weight among obese individuals after behavioral weight loss may have a similar impact in patients who undergo bariatric surgery. Additionally, no studies have examined the relationship between changes in dietary variety and food cravings, and how these factors may be related to weight loss outcomes in any population.

Primary Objectives:

To examine by surgery type(Roux-En-Y gastric bypass [RYGB], laparoscopic adjustable gastric banding [LAGB], vertical sleeve gastrectomy [VSG])

1. changes in dietary variety from pre- to post-bariatric surgery at 3, 6, and 12-months
2. changes in variety of high-energy-dense foods and changes in cravings of high-energy-dense foods at 3, 6, and 12 months and
3. changes in variety of high-energy-dense and low-energy-dense foods and changes in energy intake and weight loss at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Bariatric surgery occurring within 3-6 months

Exclusion Criteria:

* Intend to move outside of the metropolitan area within the time frame of the investigation.
* Are pregnant, lactating, less than 6 months post-partum, or plan to become pregnant during the time frame of the investigation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bariatric Surgery Patients associated with the University of Tennessee Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2011-06 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diet | 0, 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, PhD, RD, PDN, Principal Investigator — University of Tennessee
Locations (1):
- Healthy Eating and Activity Laboratory, Knoxville, Tennessee, United States

REFERENCES:
- See also: This is the website for the Healthy Eating and Activity Laboratory (HEAL), where this program is being conducted.) — http://heal.utk.edu/